CLINICAL TRIAL: NCT02320292
Title: The Asymptomatic Follicular Lymphoma (AFL) Trial: A Phase III Study of Single-Agent Rituximab Immunotherapy Versus Zevalin Radioimmunotherapy for Patients With New, Untreated Follicular Lymphoma Who Are Candidates for Observation
Brief Title: Rituximab With or Without Yttrium Y-90 Ibritumomab Tiuxetan in Treating Patients With Untreated Follicular Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: drug supply issues
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS138D; NCI-2014-02476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LS138D (Other: Mayo Clinic in Rochester); 14-003066 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Results first posted 2023-07-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2023-11

CONDITIONS: Ann Arbor Stage I Grade 1 Follicular Lymphoma; Ann Arbor Stage I Grade 2 Follicular Lymphoma; Ann Arbor Stage II Grade 1 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 1 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 2 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 2 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma
MeSH Terms: interventions — Rituximab; CT-P10; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (rituximab) (Active Comparator): Patients receive rituximab IV on days 1, 8, 15, and 22.
  Interventions: Other: Quality-of-Life Assessment; Biological: Rituximab
- Arm B (rituximab, yttrium Y-90 ibritumomab tiuxetan) (Experimental): Patients receive rituximab IV on days 1 and 8 and yttrium Y-90 ibritumomab tiuxetan over 10 minutes on day 8.
  Interventions: Other: Quality-of-Life Assessment; Biological: Rituximab; Radiation: Yttrium Y-90 Ibritumomab Tiuxetan

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Radiation: Yttrium Y-90 Ibritumomab Tiuxetan — Given IV
  Other Names: IDEC-Y2B8; IDEC-Y2B8 monoclonal antibody; Y 90 Ibritumomab Tiuxetan; Y 90 Zevalin; Yttrium Y 90 Ibritumomab Tiuxetan; yttrium Y90 ibritumomab tiuxetan
  Arms: Arm B (rituximab, yttrium Y-90 ibritumomab tiuxetan)

SUMMARY:
This phase III trial studies rituximab and yttrium Y-90 ibritumomab tiuxetan to see how well they work compared to rituximab alone in treating patients with untreated follicular lymphoma. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radioactive substances linked to monoclonal antibodies can bind to cancer cells and give off radiation which may help kill cancer cells. It is not yet known whether rituximab works better with or without yttrium Y-90 ibritumomab tiuxetan in treating follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Test the hypothesis that a single dose of Zevalin (yttrium Y-90 ibritumomab tiuxetan) rituximab immunotherapy (RIT) will increase the complete remission (CR) rate over that achieved with standard rituximab in patients with untreated asymptomatic follicular lymphoma (FL).

SECONDARY OBJECTIVES:

I. Test the hypothesis that Zevalin RIT will improve progression-free survival. II. Test the hypothesis that Zevalin RIT will improve time to next (any) therapy and time to next chemotherapy.

CORRELATIVE RESEARCH OBJECTIVES:

I. Study the incidence of exon 2 B-cell leukemia/lymphoma 2 protein (bcl2) mutations in patients with asymptomatic follicular lymphoma (AFL).

II. Measure regulatory T cells (Tregs) and tissue monocytes in on-study FL tumor tissue.

III. Measure serum cytokines and vitamin D at on study and month 6. IV. Evaluate beta-2 microglobulin plus lactate dehydrogenase (LDH) score as a prognostic factor.

V. Measure absolute lymphocyte count (ALC), absolute monocyte count (AMC), and ALC/AMC ratio at on study and after treatment.

VI. Compare quality of life as measured by the Functional Assessment of Cancer Therapy (FACT)-Lymphoma (Lym) between arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive rituximab intravenously (IV) on days 1, 8, 15, and 22.

ARM B: Patients receive rituximab IV on days 1 and 8 and yttrium Y-90 ibritumomab tiuxetan over 10 minutes on day 8.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, 18, 24, 30, 36, 48, and 60 months and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of follicular lymphoma grades I, II diagnosed within 12 months (365 days) prior to registration; NOTE: the day of biopsy should be used as day 1 of diagnosis for this calculation
* Stage I, II, III, or IV disease; NOTE: stage I disease are eligible only if the disease is not amenable to external beam radiation therapy
* No indication for chemotherapy; candidate for observation
* Measurable disease by tumor imaging with at least one lesion >= 1.5 cm in at least one dimension
* Previously untreated; NOTE: this includes any chemotherapy or immunotherapy or RIT; patients who received corticosteroids for diseases other than lymphoma are eligible as long as prednisone dose is =< 10 mg/day
* Low tumor burden as defined by Groupe d'Etudes des Lymphomes Folliculaires (GELF) criteria (2):

  * No tumor mass (nodal or extranodal) >= 7 cm in one dimension on computed tomography (CT)
  * Fewer than 3 (2 or less) nodal masses > 3 cm
  * No systemic or B symptoms
  * No splenomegaly greater than 16 cm by CT scan
  * No risk of organ compression - ureteral, orbital, neurological, gastrointestinal
  * No leukemic phase (> 5.0 x 10^9/L circulating FL cells in the blood as detected by complete blood count [CBC] with differential and smear)
  * No cytopenias - absolute neutrophil count (ANC) < 1000 or platelets < 100,000
* Meet standard criteria for RIT:

  * < 25% marrow involvement with FL
  * No evidence of myelodysplasia
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3 obtained =< 28 days prior to registration
* Platelet count >= 100,000/mm^3 =< 28 days prior to registration
* Hemoglobin > 10.0 g/dL =< 28 days prior to registration
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN, the direct bilirubin must be =< ULN =< 28 days prior to registration
* Alkaline phosphatase =< 3 x ULN =< 28 days prior to registration
* Aspartate transaminase (AST) =< 3 x ULN
* Creatinine =< 2 x ULN =< 28 days prior to registration
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to travel to a radioimmunotherapy site for Zevalin, if necessary
* Willing to return to the enrolling institution for follow-up (during the Active Monitoring Phase of the study); Note: during the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide blood samples at baseline for correlative research purposes and tissue for central pathology review
* < 25% bone marrow involvement of cellular marrow with lymphoma as determined by bilateral bone marrow aspirate and biopsy; NOTE: the percent involvement should be estimated by the hematopathologist using all of the biopsy material
* Has insurance coverage or is willing to pay for protocol therapy (rituximab x 4 or Zevalin x 1)

Exclusion Criteria:

* Any of the following because this study involves an agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception for at least three months after completing study treatment
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: These patients are excluded because it is unknown what effects prolonged B-cell depletion will have on these patient's immune system
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent that would be considered as a treatment for the lymphoma
* Active other malignancy requiring treatment that would interfere with the assessments of response of the lymphoma to protocol treatment and would interfere with follow-up assessments through year 5
* Presence of central nervous system (CNS) lymphoma
* Known to have lymphoma related to HIV or acquired immune deficiency syndrome (AIDS)
* Abnormal renal function (serum creatinine > 2 x ULN)
* Received prior external beam radiation therapy for another reason to > 25% of active bone marrow
* Serious non-malignant disease such as active infection or other condition which in the opinion of the investigator would compromise other protocol objectives
* Major surgery other than diagnostic surgery =< 4 weeks prior to registration
* Any evidence of myelodysplastic syndrome or marrow chromosomal changes suggesting myelodysplasia (-7, -5 etc)
* Corticosteroid therapy at the time the patient enters the protocol; NOTE: patients using prednisone or its equivalent for adrenal failure or using =< 10 mg of prednisone/day for other benign causes are accepted
* Follicular grades IIIA or IIIB are not eligible
* Marrow cellularity =< 15% (as determined on all bone marrow samples)
* Seropositive for or active viral infection with hepatitis B virus (HBV):

  * Hepatitis B surface antigen (HBsAg) positive
  * HBsAg negative, anti-hepatitis B surface antibody (HBs) positive and/or anti-hepatitis B core antibody (HBc) positive and detectable viral deoxyribonucleic acid (DNA)

Notes:

* Subjects who are HBsAg negative, anti-HBs positive, and/or anti-HBc positive, but viral DNA negative are eligible
* Subjects who are seropositive because of HBV vaccination are eligible (HBV surface antibody positive, HBV core antibody negative, and HBV surface antigen negative)

  * Active infection with hepatitis C virus (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Rituximab): Patients receive rituximab IV on days 1, 8, 15, and 22.> > Quality-of-Life Assessment: Ancillary studies>
  > Rituximab: Given IV
- Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan): Patients receive rituximab IV on days 1 and 8 and yttrium Y-90 ibritumomab tiuxetan over 10 minutes on day 8.>
  > Quality-of-Life Assessment: Ancillary studies>
  > Rituximab: Given IV>
  > Yttrium Y-90 Ibritumomab Tiuxetan: Given IV
Period: Overall Study
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.0 [37.0 to 84.0] | 59.0 [27.0 to 69.0] | 60.5 [27.0 to 84.0]
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 0 | 1 | 1
  30-39 | 1 | 0 | 1
  40-49 | 0 | 3 | 3
  50-59 | 4 | 1 | 5
  60-69 | 3 | 5 | 8
  70+ | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Beta-2 Microglobulin [Count of Participants; unit: Participants]
  Normal | 7 | 7 | 14
  Abnormal | 3 | 3 | 6
Time from Diagnosis to Registration [Count of Participants; unit: Participants]
  < 3 months | 8 | 7 | 15
  3-12 months | 2 | 3 | 5
Lactate Dehydrongenase [Count of Participants; unit: Participants]
  Normal | 8 | 10 | 18
  Abnormal | 2 | 0 | 2
NHL Type [Count of Participants; unit: Participants] — An indolent (slow-growing) type of non-Hodgkin lymphoma marked by enlarged lymph nodes and a mix of large cells and small cells that have cleaved (u-shaped) nuclei. Grade 1 is better, Grade 2 is worse.
  Participants
    Follicular Lymp Grade 1 | 4 | 2 | 6
    Follicular Lymp Grade 2 | 6 | 8 | 14
FLIPI2 score [Count of Participants; unit: Participants]
  Low Risk | 4 | 2 | 6
  Intermediate Risk | 6 | 6 | 12
  High Risk | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate at the 6-month Disease Assessment
Description: Will be compared between the two arms. The percentage of patients in each response category (e.g., CR, partial remission, stable disease, relapse/progressive disease) will also be tabulated by arm. The proportion of patients who have a CR at 6 months will be evaluated and compared between the two treatment regimens using a two-sided alpha=0.05 continuity corrected Cochran-Mantel-Haenszel test with stratification factors.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan)
Number analyzed (Participants) | 10 | 10
Participants
  CR | 3 | 6
  PR | 6 | 2
  SD | 1 | 2

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The distribution of progression-free survival time will be estimated using the method of Kaplan-Meier within each arm and compared between the arms using a logrank test. The progression-free survival rates at 3 years and 5 years will be estimated in each arm.
Time Frame: Time from registration to the earliest date documentation of disease progression or death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan)
Number analyzed (Participants) | 10 | 10
months | NA [23.9 to NA] — Not enough events to calculate median PFS | 29.9 [25.6 to NA] — Not enough events to calculate median PFS

3. Secondary Outcome: Time to Any Therapy (TTNT)
Description: The distribution of time to any therapy will be estimated using the method of Kaplan-Meier within each arm and compared between the arms using a log-rank test. The percentage of patients free of any therapy at 3 years and 5 years will be estimated in each arm.
Time Frame: Time from registration to the date of initiation of any treatment for follicular lymphoma, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A (Rituximab): Patients receive rituximab IV on days 1, 8, 15, and 22. >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Rituximab: Given IV
- Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan): Patients receive rituximab IV on days 1 and 8 and yttrium Y-90 ibritumomab tiuxetan over 10 minutes on day 8.
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Rituximab: Given IV
  >
  > Yttrium Y-90 Ibritumomab Tiuxetan: Given IV
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan)
Number analyzed (Participants) | 10 | 10
months | NA [47.6 to NA] — Not enough events to calculate median TTNT | 59.6 [36.1 to NA] — Not enough events to calculate median TTNT

4. Secondary Outcome: Time to Chemotherapy (TTC)
Description: The distribution of time to chemotherapy will be estimated using the method of Kaplan-Meier within each arm and compared between the arms using a log-rank test. The percentage of patients free of chemotherapy at 3 years and 5 years will be estimated in each arm.
Time Frame: Time from registration to the date of initiation of chemotherapy for follicular lymphoma, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan)
Number analyzed (Participants) | 10 | 10
months | NA [NA to NA] — Not enough events to calculate median TTC | NA [59.6 to NA] — Not enough events to calculate median TTC

5. Secondary Outcome: Incidence of Adverse Events
Description: Assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Rates of individual adverse events (grade 3 and higher) will be compared between arms using a Fisher's exact test.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan)
Number analyzed (Participants) | 10 | 10
Participants
  Grade 3+ Adverse Event | 0 | 5
  Grade 4+ Adverse Event | 0 | 1
  Grade 3+ Hem Adverse Event | 0 | 5
  Grade 4+ Hem Adverse Event | 0 | 1

6. Other Pre Specified Outcome: Incidence of Exon 2 bcl2 Mutations
Description: Will be evaluated in each arm independently and may also be compared between the two arms. Values may be investigated with respect to response (CR vs. less than CR) chi-square tests. Relationship with time to event measures (PFS, TTNT, TTC) will be evaluated using Kaplan-Meier methods and log-rank statistics (categorical measures).
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Quantification of Tissue Tregs and Tissue Monocytes on Study Tumor Biopsies
Description: Will be evaluated in each arm independently and may also be compared between the two arms. Values may be investigated with respect to response (CR vs. less than CR) chi-square tests. Relationship with time to event measures (PFS, TTNT, TTC) will be evaluated using Kaplan-Meier methods and log-rank statistics (categorical measures). For values collected at more than one time point, changes over time will be evaluated using paired-t-tests.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Serum Cytokines
Description: Each cytokine will be evaluated in reference to normal controls and levels will be categorized as normal, elevated, or suppressed. Will be evaluated in each arm independently and may also be compared between the two arms. Values may be investigated with respect to response (CR vs. less than CR) chi-square tests. Relationship with time to event measures (PFS, TTNT, TTC) will be evaluated using Kaplan-Meier methods and log-rank statistics (categorical measures). For values collected at more than one time point, changes over time will be evaluated using paired-t-tests.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Vitamin D
Description: Vitamin D level will be categorized as normal (sufficient) vs. abnormal (insufficient). Will be evaluated in each arm independently and may also be compared between the two arms. Values may be investigated with respect to response (CR vs. less than CR) chi-square tests. Relationship with time to event measures (PFS, TTNT, TTC) will be evaluated using Kaplan-Meier methods and log-rank statistics (categorical measures). For values collected at more than one time point, changes over time will be evaluated using paired-t-tests.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Beta-2 Microglobulin (B2m) Plus LDH Score
Description: Will be categorized at baseline as low risk (both factors =< 150% ULN), intermediate risk (one factor =< 150% IULN and the other factor > 150% ULN), or high risk (both factors > 150% IULN). The prognostic value of B2m plus LDH score in relation to PFS will be evaluated using Kaplan-Meier methods and log-rank statistics. Will be evaluated in each arm independently and may also be compared between the two arms.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Absolute Lymphocyte Count (ALC)
Description: Both the absolute and relative change will be summarized for each measure. Will be evaluated in each arm independently and may also be compared between the two arms. Values may be investigated with respect to response (CR vs. less than CR) chi-square tests. Relationship with time to event measures (PFS, TTNT, TTC) will be evaluated using Kaplan-Meier methods and log-rank statistics (categorical measures). For values collected at more than one time point, changes over time will be evaluated using paired-t-tests.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Absolute Monocyte Count (AMC) Ratio
Description: as for outcome 11
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in ALC/AMC Ratio
Description: as for outcome 11
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Quality of Life (QOL)
Description: As assessed by Functional Assessment of Cancer Therapy (FACT). Mean FACT will be graphically presented by arm using a mean plot with standard deviation error bars including all available data with patients according to the randomized treatment assignment. Baseline characteristics will be compared between arms within the subject of patients who provide QOL data at one or more time points using t-tests for continuous variables and chi-squared tests for categorical variables.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Arm A (Rituximab) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 1/10 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Rituximab) (N=10) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan) (N=10)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Rituximab) (N=10) | Arm B (Rituximab, Yttrium Y-90 Ibritumomab Tiuxetan) (N=10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Fatigue (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 6 (6)
Platelet count decreased (Investigations) | 0 (0) | 6 (6)
White blood cell decreased (Investigations) | 0 (0) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02320292/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT02320292/ICF_001.pdf